CLINICAL TRIAL: NCT01791504
Title: A Clinical Investigation for a Randomized Study Comparing Standard Wound Closure Technique With Drains (Control) to Standard Wound Closure Techniques Plus TissuGlu® and No Drains (Test) During Abdominoplasty
Brief Title: Clinical Trial Comparing Standard Wound Closure Techniques Versus TissuGlu® Surgical Adhesive
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-100-0085
Record Dates: First submitted 2012-12-06; First posted 2013-02-15 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Disorder of Skin and/or Subcutaneous Tissue of Trunk
Keywords: Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TissuGlu Surgical Adhesive (Experimental): Standard wound closure techniques plus TissuGlu and no drains.
  Interventions: Device: TissuGlu Surgical Adhesive
- Control - Standard of Care (No Intervention): Standard wound closure techniques with drains.

INTERVENTIONS:
Device: TissuGlu Surgical Adhesive — Standard Wound Closure Techniques Plus TissuGlu and no drains.
  Arms: TissuGlu Surgical Adhesive

SUMMARY:
The purpose of this study is to determine if TissuGlu® Surgical Adhesive is safe and effective alternative to drains(standard of care) for fluid management following abdominoplasty. It is hypothesized that the use of the Cohera device will facilitate reduction or closure of dead space when applied to planar surfaces created during an abdominoplasty procedure.

DETAILED DESCRIPTION:
The Cohera TissuGlu® study is a pivotal, prospective clinical investigation for a randomized, controlled, multicenter non-inferiority study comparing standard wound closure technique with drains (control) to standard wound closure techniques plus TissuGlu® and no drains (test) during abdominoplasty. TissuGlu® will be applied to the test group prior to standard closure of the abdominal flap thereby eliminating the deadspace between the fascia and the flap. No closed suction drains will be inserted in the test group. The control group will receive closed suction drains per the standard of care. It is hypothesized that the elimination of deadspace in the wound in the test group will prevent post-surgical fluid from developing and causing seroma and that the number of invasive treatments related to aspirations in the test group will not be inferior to the management and removal of drains and aspirations for seroma in the control group. The study will be conducted with 130 patients (65 test, 65 control) at up to 5 sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age
* Provide signed and dated informed consent form
* Willing to comply with all study procedures, schedules and be available for the follow-up evaluations for the duration of the study
* Willing to follow instructions for incision and drain care, and follow guidelines related to resumption of daily activities
* Agree not to schedule any additional elective surgical procedures that involve an incision until their participation in the study is complete
* In good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history, and review of recent concomitant medications
* Requiring at least one full thickness surgical incision of at least 20cm in length as part of elective abdominoplasty
* ≤ ASA2 - American Society of Anesthesiologists Physical Classification System (2=subject with mild systemic disease)
* Have a Body Mass Index (BMI) ≤ 28

Exclusion Criteria:

* Pregnancy or lactation
* Previous abdominoplasty
* Prior bariatric or weight loss surgery
* Lost ≥ 15% of maximum lifetime bodyweight (excluding pregnancy weight gain)
* Known medical condition that results in compromised blood supply to tissues
* Have known or suspected allergy or sensitivity to any test materials or reagents
* Have severe co-morbid conditions (e.g., heart disease)
* Are currently a smoker or have smoked within 30 days of prescreening as determined by nicotine test
* Any condition known to effect wound healing, such as collagen vascular disease
* Be known to have a blood clotting disorder and/or be willing to discontinue anti-coagulation therapy including aspirin
* Diagnosis of diabetes with current medical treatment
* Receiving antibiotic therapy for pre-existing condition or infection
* Have known personal or family history of keloid formation or hypertrophic scarring
* Currently taking systemic steroids or immunosuppressive agents
* Undergoing concurrent adjacent or congruent Liposuction agents
* Use of pain pumps after the abdominoplasty procedure
* Concurrent use of fibrin sealants or other internal wound care devices
* Concurrent hernia repair greater than 6 cm and/or requiring the use of mesh
* Mini abdominoplasty (abdominoplasty without umbilical transposition)
* Be participating in any current clinical trial or have participated in any clinical trial within 30 days of enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Post-Operative Invasive Treatments | 90 Days
  Number of Post-Operative Invasive Treatments, where Invasive Treatment is defined as one of the following events:
  * Removal of an in-dwelling drain;
  * Needle aspiration to remove fluid from a clinically-diagnosed palpable seroma;
  * Invasive action to the drain or drain wound such as repositioning or re-attaching the drain retention sutures;
  * Reinsertion of a drain

SECONDARY OUTCOMES:
Secondary Outcome Measures | 90 Day
  • Cumulative drain volume, aspiration volume, and total wound drainage (drain volume + aspiration volume)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hunstad, MD, Principal Investigator — The Hunstad Kortesis Center for Cosmetic Plastic Surgery and MedSpa
Locations (1):
- The Hunstad Kortesis Center for Cosmetic Plastic Surgery and MedSpa, Huntersville, North Carolina, United States